CLINICAL TRIAL: NCT05826938
Title: Can Virtual Reality Technology Improve the Patient Experience in Oocyte Retrieval?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Consultant, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Virtual Reality-project
Record Dates: First submitted 2023-03-08; First posted 2023-04-24 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Infertility, Female
Keywords: Infertility; Virtual reality
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): The intervention group receives stimuli in the form of Virtual Reality technology before and during oocyte retrieval. In addition, patients receive standard treatment
  Interventions: Device: Virtual reality technology
- Control (No Intervention): The control group, does not receive stimuli in the form of Virtual Reality technology, but only the standard treatment

INTERVENTIONS:
Device: Virtual reality technology — Participants who are randomized to group 1 will receive the Virtual Reality glasses on the day of oocyte retrieval in the recovery room. The participant chooses which animation she wants to experience.
  Arms: Virtual reality

SUMMARY:
A non-pharmacological, non-blinded, randomized cohort study that will investigate the effect of Virtual Reality technology on the patient experience during oocyte retrieval.

The primary objective of the trial is to investigate the impact of Virtual Reality technology on the patient experience

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing oocyte retrieval
* Understanding and speaking Danish

Exclusion Criteria:

* Previous participation in the trial
* Acupuncture as pain relief during oocyte retrieval

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-13 (Estimated)

PRIMARY OUTCOMES:
Questionnaires regarding impact on patient experience | 30-60 minutes
  The impact of Virtual Reality technology on the patient experience during oocyte retrieval through questionnaires.
  A visual analog scale (VAS) from 1-10 will be used for this measurement.

SECONDARY OUTCOMES:
Questionnaires reagarding the impact on the consumption of analgesic medication | 30-60 minutes
  The effect of Virtual Reality technology on the consumption of analgesic medication.
  A visual analog scale (VAS) from 1-10 will be used for this measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Skive, Skive Regional Hospital, Skive, Denmark